CLINICAL TRIAL: NCT00736619
Title: Phase I Study of Weekly Nanoparticle Albumin-Bound Paclitaxel (Abraxane) + Weekly Cetuximab + Radiation Therapy (IMRT, Intensity-Modulated Radiation Therapy) in Patients With Stage III-IVB Head and Neck Squamous Cell Carcinoma (HNSCC)
Brief Title: Weekly Nanoparticle Albumin-Bound Paclitaxel (Abraxane) + Weekly Cetuximab + Radiation Therapy (IMRT, Intensity-Modulated Radiation Therapy) in Patients With Stage III-IVB Head and Neck Squamous Cell Carcinoma (HNSCC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Celgene Corporation (Industry); National Comprehensive Cancer Network (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-084
Record Dates: First submitted 2008-08-15; First posted 2008-08-18 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: HEAD & NECK Cancer
Keywords: MAB C225(CETUXIMAB)(ANTI-EGFR); TAXOL (PACLITAXEL); Radiation Therapy; 08-084
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Cetuximab; Radiotherapy, Intensity-Modulated; Albumin-Bound Paclitaxel

ARMS (1):
- 1 (Experimental): Cetuximab loading dose, 400 mg/m2 intravenously (IV) IMRT, 1 fraction/day, up to total of approximately 70 Gy, over approximately 33 treatment days
  * Cetuximab 250 mg/m2 weekly IV X 7 weeks
  * Albumin-bound paclitaxel (Abraxane®) weekly IV X 7 weeks, according to dose escalation scheme
  Interventions: Other: Cetuximab, IMRT, Albumin-bound paclitaxel (Abraxane®)

INTERVENTIONS:
Other: Cetuximab, IMRT, Albumin-bound paclitaxel (Abraxane®) — All patients will receive standard treatment with definitive radiation therapy (IMRT, intensity-modulated radiation therapy) administered concurrently with cetuximab (400 mg/m2 intravenous loading dose one week prior to radiation therapy, followed by 250 mg/m2 weekly intravenous infusions). To explore different dose levels of nanoparticle albumin-bound paclitaxel (Abraxane®) given intravenously weekly with the standard regimen of weekly cetuximab + daily radiation therapy.
  The total number of planned cetuximab infusions is 8 (loading dose, plus 7 weekly infusions concurrent with radiation therapy). The total number of planned albumin-bound paclitaxel infusions is 7 (all concurrent with radiotherapy). Five dose levels of weekly intravenous (IV) albumin-bound paclitaxel will be explored.

SUMMARY:
For patients with this type of cancer, one standard treatment option is cetuximab (Erbitux®) + radiation. We wish to study the addition of albumin-bound paclitaxel (Abraxane®) to this standard regimen of cetuximab + radiation. Albumin-bound paclitaxel and cetuximab both are chemotherapy drugs which are administered by vein.

Previous studies have shown that albumin-bound paclitaxel can kill head and neck cancer cells when given alone or in combination with chemotherapy. The purpose of this study is to establish a safe dose range of albumin-bound paclitaxel given in combination with cetuximab and radiation therapy. The investigators want to find out what effects, good and/or bad, the albumin-bound paclitaxel has on you and your head and neck cancer.

ELIGIBILITY:
Inclusion Criteria:

* Locally and/or regionally advanced head and neck squamous cell carcinoma (AJCC Stage III-IVB)
* Karnofsky performance status ≥ or = to 70%
* Adequate bone marrow function: absolute neutrophil count ≥ or = to 1,500/μl, platelets ≥ or = to 100,000/μl, hemoglobin ≥ or = to 9 gm/dl
* Adequate hepatic function:

Total Bilirubin ≤ or = to institutional upper limit of normal (ULN) AST and ALT and Alkaline Phosphatase must be within the range allowing for eligibility. In determining eligibility the more abnormal of the two values (AST or ALT) should be used

* Patients must have adequate renal function: serum creatinine ≤ 1.5 mg/dl or estimated creatinine clearance of ≥ 45 ml/min by Cockcroft and Gault method
* Men and women of childbearing potential must be willing to consent to using effective contraception while on treatment and for at least 3 months thereafter
* Women of childbearing potential must have a negative pregnancy test
* Patients must have ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Other active malignancy, other than indolent malignancies which the investigator determines are unlikely to interfere with treatment or efficacy analysis. For example, patients with non-melanoma skin cancer, in situ carcinoma of the cervix, or prostate cancer within the no current biochemical (PSA) or radiologic evidence of disease may enroll
* Prior radiation therapy for head and neck cancer
* Patients with multifocal peripheral sensory alterations or paresthesias (including tingling) interfering with function, per patient report (example: activities of daily living)
* Inability to comply with study and/or follow-up procedures
* Women who are pregnant or lactating
* Serious concomitant medical disorders (for example, active infection, uncontrolled seizure disorder, unstable angina, auto-immune connective tissue disease) that, in the opinion of the investigator, would compromise the safety of the patient or compromise the patient's ability to complete the study
* History of severe infusion reaction to a monoclonal antibody
* Patients with nasopharyngeal carcinoma are not eligible

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-08; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
To establish the phase II recommended dose of weekly intravenous albumin-bound paclitaxel (Abraxane®) given concurrently with weekly cetuximab + definitive radiation therapy (IMRT) for patients with HNSCC. | conclusion of study

SECONDARY OUTCOMES:
To establish the safety and tolerability of weekly albumin-bound paclitaxel + cetuximab + RT for patients with HNSCC. | conclusion of study

CONTACTS AND LOCATIONS:
Overall Officials: David Pfister, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memorial Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center, Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering at Mercy Medical Center, Rockville Centre, New York
  - Memoral Sloan Kettering Cancer Center@Phelps, Sleepy Hollow, New York

REFERENCES:
- [Derived] Fury MG, Sherman EJ, Rao SS, Wolden S, Smith-Marrone S, Mueller B, Ng KK, Dutta PR, Gelblum DY, Lee JL, Shen R, Kurz S, Katabi N, Haque S, Lee NY, Pfister DG. Phase I study of weekly nab-paclitaxel + weekly cetuximab + intensity-modulated radiation therapy (IMRT) in patients with stage III-IVB head and neck squamous cell carcinoma (HNSCC). Ann Oncol. 2014 Mar;25(3):689-694. doi: 10.1093/annonc/mdt579. Epub 2014 Feb 3. PMID 24496920
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org